CLINICAL TRIAL: NCT06979687
Title: Knotless Barbed Suture Closure of the Uterus at Caesarean Section
Status: Completed | Type: Observational
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24/022
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-01

CONDITIONS: Caesarean Section; Caesarean Section; Infection
Keywords: Knotless barbed suture; caesarean section; caesarean delivery; caesarean birth
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1 (Elective Caesareans undertaken using knotless barbed suture): Elective caesareans undertaken using knotless barbed sutures. This included all cases without exception on the CI's regular operating list from January 2023 (after a positive trial period which resulted in this becoming the standard for the CI). n290.
  Interventions: Procedure: knotless barbed suture closure of the hysterotomy at caesarean section
- Group 2 (Elective caesarean sections on a number of consultant lists using standard sutures SS): May-August 2024 all cases on the respective lists n215
  Interventions: Procedure: Standard 2 layer closure of caesarean hysterotomy using 910 polyglactin suture (SS)
- Group 3 (Emergency caesarean deliveries when KBS was used for closure of the hysterotomy): Emergency caesarean deliveries (category 1-3 urgency - all except elective) using KBS January 2023-December 2024. n 107.
  Interventions: Procedure: knotless barbed suture closure of the hysterotomy at caesarean section
- Group 4 (Emergency caesarean deliveries employing Standard sutures for closure of the hysterotomy): All non-cat 4 CS using SS (May-August 2024) n 345
  Interventions: Procedure: Standard 2 layer closure of caesarean hysterotomy using 910 polyglactin suture (SS)
- Group 5 (comprising all cases in group 1 and group 3): All the KBS caesarean deliveries n 397
  Interventions: Procedure: knotless barbed suture closure of the hysterotomy at caesarean section
- Group 6 (comprising group 2 and group 4): All the SS cases n560
  Interventions: Procedure: Standard 2 layer closure of caesarean hysterotomy using 910 polyglactin suture (SS)

INTERVENTIONS:
Procedure: knotless barbed suture closure of the hysterotomy at caesarean section — Use of Medtronic V-loc 180 suture (VL) for a 2 layer closure of the caesarean hysterotomy rather than the standard 2 layer closure using the 910 polyglactin suture (SS).
  Groups: Group 1 (Elective Caesareans undertaken using knotless barbed suture); Group 3 (Emergency caesarean deliveries when KBS was used for closure of the hysterotomy); Group 5 (comprising all cases in group 1 and group 3)
Procedure: Standard 2 layer closure of caesarean hysterotomy using 910 polyglactin suture (SS) — Standard 2 layer closure using the 910 polyglactin suture (SS)
  Groups: Group 2 (Elective caesarean sections on a number of consultant lists using standard sutures SS); Group 4 (Emergency caesarean deliveries employing Standard sutures for closure of the hysterotomy); Group 6 (comprising group 2 and group 4)

SUMMARY:
Caesarean section (CS) is an increasingly common mode of delivery. The way in which this operation is carried out is important as it affects millions of women each. In recent years use of a 'self-retaining' suture or thread for closure of the uterine closure has become a recognised approach with a proven safety record. These sutures are known as knotless barbed sutures (KBS) as the unidirectional barbs on the surface of the suture hold the suture in the tissue without the need for knots. These sutures can be used instead of the usual 'smooth' suture which requires knots at the angles. There are high-level level data that CS are quicker and on average need fewer additional stitches to control blood loss when KBS are used. There is additional evidence of a potential reduction in problems with healing of the uterus with KBS, it is thought that this might lead to a lower risk of problems in repeat CS as the chance of the placenta implanting into the scar might be lower. At present this evidence is based on ultrasound surveillance of scar appearance which is an indirect measure. The real risk difference will need to be explored with the examination of real world outcomes over the coming years.

There is currently no published data on KBS for uterine closure at caesarean from the UK. This cohort, although retrospective, is adequately controlled, shows excellent outcomes and signals a potential marked reduction in infectious morbidity. This potentially means a better patient experience as well as a large cost saving because of reduced re-admission rates. These data were collected as part of a service improvement project but the generalisable nature of our findings mean the finding are research and should be published.

DETAILED DESCRIPTION:
Caesarean section (CS) is one of the most commonly performed operations worldwide and the prevalence is increasing1. There are perioperative complications including neonatal morbidity and, on the maternal side, haemorrhage, infection and organ injury2. Furthermore, there are implications for future pregnancies, the risks of which rise with each successive caesarean3. Closure of the lower segment hysterotomy at CS is most commonly affected using a 2-layer approach employing braided absorbable sutures such as Vicryl (polyglactin 910)4. Closure is with a continuous suturing technique and the tension of the closure is maintained manually until the suture is secured with knots at the angles. Knotless barbed suture (KBS) closure of the caesarean hysterotomy remains a novel technique that is not yet widely employed. These sutures, first invented in 1964, were approved by the FDA in 2004 and were first used in a clinical trial in 20075. Barbed sutures anchor themselves within the tissue, as barbs on the suture resist backward movement through the tissue. They offer even tension over the length of the hysterotomy and are cut flush with the uterus without the need for anchoring knots.

A systematic review and meta-analysis of randomised control trials (n460) on KBS compared with 'smooth' sutures at elective CS found that operative times were lower and the need for additional haemostatic sutures was lower6. There was a trend towards lower blood loss and no difference in operative morbidity. Some trials, some of which are ongoing, have examined whether there is a difference in lower segment residual myometrial thickness (RMT) after KBS and whether there is a difference in the incidence of scar niche7. These outcomes, respectively, are offered as potential proxy measures for uterine rupture risk and praevia or PAS risk. The results of these trials, as per their proxy outcomes, have been encouraging. This trial offers the first data on KBS at CS in UK practise.

Methods:

This single-centre retrospective cohort study in a tertiary care hospital in Northern England including caesarean deliveries from November 2022 to October 2024 - a 24 month period. The cohorts are women who had a Medtronic's V-loc 180 absorbable device (KBS) and women who had 2 layer vicryl (polyglactin 910) uterine closure i.e. smooth suture (SS).

Data was collected prospectively using a Microsoft Excel™ spreadsheet by the lead clinician (HS) as part of a quality improvement project and data was cross-referenced with patient records using Clevermed badgernotes ™ maternity system data records. Baseline characteristics reported are: patient age at delivery, parity, number of previous caesarean sections, BMI at booking, additional intraoperative interventions, birth-weight, indication for, and category of, caesarean, mode of anaesthesia, grade of operator and whether a consultant was present if not the primary surgeon (Table 1). The pre-specified outcome was blood loss. The pre-specified secondary outcomes were operating time, infection rates, readmission, unplanned outpatient attendance, and other complications.

Women were grouped for comparison as follows: group 1, n290 elective CS undertaken using KBS (November 2022-December 2024); group 2 - n215 Elective caesareans undertaken on a number of consultant lists using SS (May-August 2024). Group 3 - n107 Emergency caesarean deliveries using KBS (January 2023-December 2024); Group 4 - n345 emergency caesarean deliveries using SS (May-August 2024). Group 5 - n397 comprises group 1 and group 3. Group 6 - n560 comprises group 2 and group 4. The plan for data analysis was pre-specified and published prior to analysis being undertaken.

The investigators report baseline characteristics and outcomes as means (SDs), or numbers and percentages. Difference in outcome by cohort is reported as relative risk with 95% CI. Multivariate analysis was used to assess correlation for inclusion of variables in binary logistic regression for adjustment of risk. Variables felt relevant were included regardless of significance of correlation, as pre-specified - for the primary outcome, across all three comparisons, the following variables were pre-selected for inclusion in adjustment of risk: BMI, birthweight, mode of anaesthesia. For the secondary outcomes pre-specified variables for adjustment of risk across all three comparisons were as follows: for operating time; BMI, additional operative interventions, number of previous caesareans, for infection rates; BMI, category of caesarean and indication, for readmission; BMI and category of caesarean, for unplanned outpatient attendances as for readmission. There was no planed adjustment for the safety outcome of other complications. Unpaired t-tests, Chi square or Fisher's exact test were used to test significance for categorical and continuous outcomes. Analysis was carried out using IBM SPSS version 24. Alpha was taken as 0.05 for the primary outcome and 0.01 for the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a caesarean section at the study hospital within the data collection period for that cohort - either with or without KBS depending on the cohort.

Exclusion Criteria:

* Not falling within the search criteria for a comparator group

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women having a caesarean section at James Cook University Hospital within the study period
Sampling Method: Non-Probability Sample
Enrollment: 957 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Post-operative infection | up to 6 weeks post-operative
  Whether antibiotics were prescribed for a surgical site infective complication.

SECONDARY OUTCOMES:
operating time | Intraoperative
  Time from knife to skin to closure of skin
Blood loss | In theatre during the operation
  Estimated or measured intraoperative blood loss (estimates are used unless blood loss is thought excessive when measuring is carried out contemporaneously)
Readmission | up to 6 weeks post-operative
  Readmission to hospital within 6 weeks post-operative for a maternal indication (not a neonatal one)
Re-attendance as an outpatient | up to 6 weeks post-operative
  Attending hospital as an outpatient for an unscheduled review

OTHER OUTCOMES:
Operative complications | Intraoperative and up to 6 weeks post-operatively
  Failure of the suture (snapping intraoperatively), organ injury (bladder, bowel, ureter), major haemorrhage (>1.5 litre loss) or other unexpected adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- James Cook University Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared via CT.gov on an excel spreadsheet without identifiable information being provided
Supporting Information: Study Protocol, SAP
Time Frame: Feb 2025
Access Criteria: Open access on CT.gov
URL: http://clinicaltrials.gov